CLINICAL TRIAL: NCT05875324
Title: The Effect of Virtual Reality on Pain, Kinesiophobia and Function in Total Knee Arthroplasty Patients
Brief Title: Effects of Virtual Reality in TKA Patients
Acronym: TKA
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Kırklareli University (Other)
Collaborators: Gazi University (Other)
Responsible Party: Principal Investigator, Ozan Gür, PT, Research Assistant, Kırklareli University
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 611
Record Dates: First submitted 2023-05-13; First posted 2023-05-25 (Actual); Last update posted 2023-05-25 (Actual); Status verified 2023-05

CONDITIONS: Knee Arthropathy
Keywords: Knee arthroplasty; VR; Exercise; Pain; Kinesiophobia; Catastrophization; Function
MeSH Terms: conditions — Motor Activity; Pain; Kinesiophobia | interventions — Exercise

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- VR Group (Experimental): The patients in the VR group were informed about the disease, the goals of post-surgical rehabilitation, the exercises, and the circumstances to be considered following TKA. On the postoperative first day, activities included sitting on the side of the bed and mobilizing in and out of the room using a walker. Patients were discharged 2.5 days after surgery. Patients were provided an exercise program for at-home practice. In addition to the exercise program, VR glasses were used before the exercises in the VR group. The second examination was performed three days after the completion of treatment.
  Interventions: Device: virtual reality application; Other: exercise
- Exercise Group (Active Comparator): Exercise group were informed about the disease, the goals of post-surgical rehabilitation, the exercises, and the circumstances to be considered following TKA. On the postoperative first day, activities included sitting on the side of the bed and mobilizing in and out of the room using a walker. Patients were discharged 2.5 days after surgery. Patients in the exercise group were provided an exercise program for at-home practice. The second examination was performed three days after the completion of treatment.
  Interventions: Other: exercise

INTERVENTIONS:
Device: virtual reality application — VR was used for 10 minutes a day in the sitting position for three weeks, twice a week, by watching a walking video before beginning the exercises. Patients were instructed to imagine themselves walking while concentrating on walking and watching the video. The patients were asked to stop watching video by removing their VR glass if they experienced discomfort such as dizziness and nausea during the VR application. They were told to continue watching the video when the discomfort was gone. In cases where similar discomforts recurred, the treatment was terminated.
  Arms: VR Group
Other: exercise — activities included sitting on the side of the bed and mobilizing in and out of the room using a walker. Patients were provided an exercise program for at-home practice.

SUMMARY:
The goal of this clinical trial] is to investigate the effects of virtual reality (VR) in patients undergoing total knee arthroplasty (TKA). The main questions it aims to answer are:

* Does VR have effects on pain, kinesiophobia, and function during the early rehabilitation period of patients who have undergone TKA
* Does VR contribute to the success of exercise treatment after TKA

All the patients included in the study were informed about the disease, the goals of post-surgical rehabilitation, the conditions to be considered after TKA and exercises. Sitting on the side of the bed and mobilization in or out of the room with a walker were provided with the postoperative 1st day exercises. The patients were discharged 2.5 days after surgery. The patients in both groups were taught an exercise program for home practice.

In addition to the exercise program, the virtual reality application was applied before the exercises to the VR group. The second evaluation was made 3 days after the end of the treatment in both patient groups.

Researchers compared VR and exercise to see if pain, kinesiophobia, pain catastrophizing, knee range of motion, function, and quality of life had changed.

ELIGIBILITY:
Inclusion Criteria:

* Being between the ages of 50 and 70
* Being female
* Having received TKA due to being at stage III or IV according to the Kellgren-Lawrence Osteoarthritis Classification
* Having sufficient eyesight
* Having kinesiophobia and pain catastrophizing

Exclusion Criteria:

* Having undergone bilateral knee arthroplasty/revision knee arthroplasty
* Vertigo or motion-sensitive nausea
* Being diagnosed with an additional neurological, rheumatological, or oncological disease
* Having a Mini Mental Test score of less than 24
* Being diagnosed with severe anxiety by a specialist physician
* Inability to complete the treatment program

Ages: 50 Years to 70 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Gender Based: Yes — It has been determined that women's proportion of knee extensors, knee flexors and knee Flexors / extensors ratio when compared with men, the ratio of the knee extender and flexor muscle groups is different in relation to the overall body muscle mass, and there are differences in functional outcomes in women and men in the early post-TKA period. It is also believed that women have more pain sensitivity than men and that pain inhibition mechanisms are less effective. Only female patients were included in this study because differences between groups and within-groups could not affect the results of the study.
Enrollment: 21 (Actual)
Dates: Start 2019-10-13 (Actual); Primary Completion 2021-08-10 (Actual); Study Completion 2021-08-10 (Actual)

PRIMARY OUTCOMES:
Kinesiophobia assessed by Tampa Kinesiophobia Scale | first day after TKA
  Kinesiophobia was evaluated by using the Tampa Kinesiophobia Scale (total score between 17-68) (higher values indicate higher kinesiophobia). The Tampa Kinesiophobia Scale includes the parameters of injury/re-injury and fear of movement; scores of 37 and above indicate the presence of high kinesiophobia (ICC: 0,806).
Kinesiophobia assessed by Tampa Kinesiophobia Scale | 4th week after TKA
  Kinesiophobia was evaluated by using the Tampa Kinesiophobia Scale (total score between 17-68) (higher values indicate higher kinesiophobia). The Tampa Kinesiophobia Scale includes the parameters of injury/re-injury and fear of movement; scores of 37 and above indicate the presence of high kinesiophobia (ICC: 0,806).

SECONDARY OUTCOMES:
knee pain assessed by Numerical Pain Rating Scale | first day after TKA
  The intensity of pain was evaluated by using the Numerical Pain Rating Scale (score between 0-10) (higher values indicate higher pain) at rest, at night and during functional tests (ICC: 0,84).
knee pain assessed by Numerical Pain Rating Scale | 4th week after TKA
  The intensity of pain was evaluated by using the Numerical Pain Rating Scale (score between 0-10) (higher values indicate higher pain) at rest, at night and during functional tests (ICC: 0,84).
pain catastrophizing assessed by Pain Catastrophizing Scale | first day after TKA
  Pain catastrophizing was evaluated by using the Pain Catastrophizing Scale (total score between 0-52) (higher values indicate higher pain catastrophizing). The scores of 30 and above taken from the Pain Catastrophizing Scale indicate the presence of high pain catastrophizing (ICC: 0,83).
pain catastrophizing assessed by Pain Catastrophizing Scale | 4th week after TKA
  Pain catastrophizing was evaluated by using the Pain Catastrophizing Scale (total score between 0-52) (higher values indicate higher pain catastrophizing). The scores of 30 and above taken from the Pain Catastrophizing Scale indicate the presence of high pain catastrophizing (ICC: 0,83).
knee range of motion assessed by universal goniometer | first day after TKA
  ROM was measured with a universal goniometer. Active flexion and extension measurements were performed while the patients were lying in the supine position (ICC: 0.81; ICC: 0.86, respectively). In the knee extension evaluation, cases where 0° could not be reached in the evaluation of knee extension were recorded as positive values, and the degrees of knee extension performed more than the initial position of 0° were recorded as negative values.
knee range of motion assessed by universal goniometer | 4th week after TKA
  ROM was measured with a universal goniometer. Active flexion and extension measurements were performed while the patients were lying in the supine position (ICC: 0.81; ICC: 0.86, respectively). In the knee extension evaluation, cases where 0° could not be reached in the evaluation of knee extension were recorded as positive values, and the degrees of knee extension performed more than 0° were recorded as negative values.
objective functional measurement assessed by functional tests | first day after TKA
  For the Five Times Sit to Stand Test (time-second), subjects were asked to rise from a standard height (43 cm) chair without armrests, five times, as fast as possible with their arms folded (ICC: 0.80).
  For the Timed Up and Go Test (time-second), subjects were asked to rise from sitting in an armchair, walk 3 meters, turn, walk back to the chair, then sit down and a walking aid if required (ICC: 0.97).
  For the Stair Climb Test (time-second), subjects were asked to ascend steps at the bottom of eight steps (15 cm high, 27.5 cm deep). Subjects could use the handrail if preferred and a walking aid if they normally used one. After a brief rest, the subject was asked to descend the stairs (ICC: 0.93).
objective functional measurement assessed by functional tests | 4th week after TKA
  For the Five Times Sit to Stand Test (time-second), subjects were asked to rise from a standard height (43 cm) chair without armrests, five times, as fast as possible with their arms folded (ICC: 0.80).
  For the Timed Up and Go Test (time-second), subjects were asked to rise from sitting in an armchair, walk 3 meters, turn, walk back to the chair, then sit down and a walking aid if required (ICC: 0.97).
  For the Stair Climb Test (time-second), subjects were asked to ascend steps at the bottom of eight steps (15 cm high, 27.5 cm deep). Subjects could use the handrail if preferred and a walking aid if they normally used one. After a brief rest, the subject was asked to descend the stairs (ICC: 0.93).
subjective functional measurement assessed by Western Ontario and McMaster Universities Osteoarthritis Index | first day after TKA
  The Western Ontario and McMaster Universities Osteoarthritis Index (WOMAC) (total score between 0-96) (higher values indicate worse function) is a disease-specific, self-administered questionnaire developed to study patients with hip or knee OA. It consists of 24 questions, grouped into 3 subscales (pain, stiffness, and physical function). In Likert scale, there are five alternative answers to every question (0=none, 1=mild, 2=moderate, 3=severe, 4=extreme). The maximum score in Likert scale scale is 20 points for pain, 8 points for stiffness, and 68 points for physical function (ICC: 0.71-0.94).
subjective functional measurement assessed by Western Ontario and McMaster Universities Osteoarthritis Index | 4th week after TKA
  The Western Ontario and McMaster Universities Osteoarthritis Index (WOMAC) (total score between 0-96) (higher values indicate worse function) is a disease-specific, self-administered questionnaire developed to study patients with hip or knee OA. It consists of 24 questions, grouped into 3 subscales (pain, stiffness, and physical function). In Likert scale, there are five alternative answers to every question (0=none, 1=mild, 2=moderate, 3=severe, 4=extreme). The maximum score in Likert scale scale is 20 points for pain, 8 points for stiffness, and 68 points for physical function (ICC: 0.71-0.94).
quality of life assessed by Short Form 36 | first day after TKA
  Quality of life was evaluated using the Short Form 36 (SF-36) quality of life scale (total score between 0-100 for each subscale) (higher values indicate better health). SF-36 consists of a total of 36 items belonging to 8 different subgroups called physical, social, emotional function, physical role, mental health, fatigue, pain, and general health. An increase in the score indicates better health, while a decrease indicates worse health (Cronbach's Alpha: 0.7324-0.7612).
quality of life assessed by Short Form 36 | 4th week after TKA
  Quality of life was evaluated using the Short Form 36 (SF-36) quality of life scale (total score between 0-100 for each subscale) (higher values indicate better health). SF-36 consists of a total of 36 items belonging to 8 different subgroups called physical, social, emotional function, physical role, mental health, fatigue, pain, and general health. An increase in the score indicates better health, while a decrease indicates worse health (Cronbach's Alpha: 0.7324-0.7612).

CONTACTS AND LOCATIONS:
Locations (1):
- Kırklareli University, Kırklareli, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: Undecided